CLINICAL TRIAL: NCT00979706
Title: Immune-based Therapy Pilot Study for the Treatment of Primary HIV Infection With the Objective to Induce a Strong Specific HIV Immune Response Able to Control Viral Replication Without Highly Active Anti-Retroviral Therapy (HAART)
Brief Title: Immune-based Therapy Pilot Study for the Treatment of Primary HIV Infection (PHI-IMD).
Acronym: PHI-IMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, MDPhD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHI-INMUNOMEDIADO
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: HIV
MeSH Terms: interventions — Antiretroviral Therapy, Highly Active; Tenofovir; Lamivudine; lopinavir-ritonavir drug combination; Immunotherapy; Cyclosporine; Granulocyte-Macrophage Colony-Stimulating Factor; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HAART (Active Comparator): Patients assigned to this arm will receive standard HAART
  Interventions: Drug: HAART
- HAART + Immunotherapy (Experimental): Patients assigned to this arm will receive HAART plus cyclosporin A during the first two months and after that will receive IFN, GM-CSF and IL-2.
  Interventions: Drug: HAART + Immunotherapy

INTERVENTIONS:
Drug: HAART — Patients assigned to this arm will receive Trizivir and kaletra. After the first 9 months of HAART, all patients will stop HAART until HIV viral load in plasma became detectable (>200 copies/mL). Then, they will re-start HAART plus low doses of IL-2 during 2 months.
  All patients will be followed-up during 1 year.
  Other Names: Viread; Epivir; Kaletra
  Arms: HAART
Drug: HAART + Immunotherapy — Patients assigned to this arm will receive Trizivir + Kaletra + cyclosporin A during the first two months. This group also will receive GM-CSF plus pegylated-interferon-alpha until HIV viral load in plasma became detectable (>200 copies/mL). Then, they will re-start HAART plus low doses of IL-2 during 2 months. At this moment they will stop HAART.
  All patients will be followed-up during 1 year.
  Other Names: Cyclosporine A; GM-CSF; Peg-IFN; Interleukin-2
  Arms: HAART + Immunotherapy

SUMMARY:
Pilot study for the treatment of primary HIV infection with the objective to induce a strong specific HIV immune response able to control viral replication without HAART.

DETAILED DESCRIPTION:
Pilot and open RCT in 20 patients with primary HIV-1 infection who were randomized to one of these two arms: 1) Control arm (A), Tenofovir +Lamivudine + Lopinavir-ritonavir (Kaletra) at standard doses for 44 weeks (W44); a short treatment interruption (TI) was performed at W36, and HAART was restarted for 8 weeks when plasma HIV-1 RNA viral load (pVL) rebounded>200 copies/mL. At W44 HAART was stopped and patients were followed for 48 additional weeks (W92). 2) Immune-based arm (B), same HAART schedule plus oral cyclosporine A (CsA)(serum levels 250-350 mcg/L) for the first 8 weeks of HAART. During the TI, patients received sc GM-CSF (250 mcg TIW) plus weekly sc pegylated-interferon a2b (Peg-INF)(1.5 mcg/kg/week). During the last 8 weeks of HAART (until W44), patients received daily sc low-dose interleukin-2 (IL-2)(0.75 MU/kg QD). The primary endpoint was pVL <1000copies/mL (<3.0 log10/mL) at 12 (W56) and at 48 (W92) weeks after stopping HAART. Sample size was calculated in order to detect a pVL difference of 1.5log10 copies/mL at 12 (W56) weeks after stopping HAART between the control and the immune-based arms with a power of 80% and a level of significance of0.05.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected patients (age 18 years or over) with primary HIV infection <90 days.
2. Giving written informed consent to participate into the study.

Exclusion Criteria:

1. Patients not accepting to start HAART. Patients wishing start HAART treatment with nevirapine or efavirenz.
2. Pregnant women or planning pregnancy.
3. Intravenous drug user or alcohol abuse.
4. Previous treatment with cyclosporin A, GM-CSF,pegylated-interferon-alpha o interleukine-2.
5. Renal or liver failure.
6. Any formal contraindication to treatment with the study drugs.
7. Patients with a history of psychiatric disorder, thyroid illness, dislipidemia requiring treatment, cardiovascular disease, arterial hypertension, or diabetes mellitus.
8. In treatment with drugs interacting with study drugs.
9. Acute infection for HTLV-I or EBV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients remaining below 5,000 copies/mL at 12 and 48 weeks after stoping HAART. | W12 y W48

SECONDARY OUTCOMES:
Adherence to treatment | W8, W24, W36, W96
CD4, CD8 | W8, W24, W36, W96
Specific HIV immune responses (CD4 and CTL) | W8, W24, W36, W96
Proportion of patients PVL (plasma viral load)<40 | W8, W24, W36, W96
Adverse events | W8, W24, W36, W96

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria Miró, MDPhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Nicolas D, Ambrosioni J, Sued O, Brunet M, Lopez-Dieguez M, Manzardo C, Aguero F, Tuset M, Plana M, Guardo AC, Mosquera MM, Munoz-Fernandez MA, Caballero M, Marcos MA, Gatell JM, de Lazzari E, Gallart T, Miro JM. Cyclosporine A in addition to standard ART during primary HIV-1 infection: pilot randomized clinical trial. J Antimicrob Chemother. 2017 Mar 1;72(3):829-836. doi: 10.1093/jac/dkw462. PMID 27999018